CLINICAL TRIAL: NCT05242900
Title: Imaging Sodium and Lymphatics in Lymphedema
Status: Active, not recruiting | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Rachelle Crescenzi, Associate Professor, University of Virginia
Other Study IDs: 302403; 1R01HL155523-01 (NIH); 202424 (Other: Vanderbilt University Medical Center)
Record Dates: First submitted 2021-12-07; First posted 2022-02-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Lymphedema of Leg; Lymphedema, Secondary; Lymphedema Related Fibrosis
Keywords: MRI; sodium; lymphedema; adipose tissue; fibrosis
MeSH Terms: conditions — Lymphedema; Neoplasm Metastasis; Fibrosis | interventions — Manual Lymphatic Drainage; Exercise

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- At-risk for lymphedema: Participants at-risk for leg lymphedema
  Interventions: Other: Standard imaging protocol
- With lymphedema: Participants with leg lymphedema
  Interventions: Other: Standard imaging protocol
- With lymphedema undergoing complete decongestive therapy (CDT): Participants with leg lymphedema undergoing routine complete decongestive therapy (CDT)
  Interventions: Procedure: Complete decongestive therapy; Other: Standard imaging protocol

INTERVENTIONS:
Procedure: Complete decongestive therapy — The investigators will identify participants undergoing clinically-indicated interventions that they are already receiving for their routine clinical management (complete decongestive physical therapy). They will make no evaluation of the efficacy of these procedures, but rather will test fundamental hypotheses regarding lymphatic clearance of tissue sodium.
  Other Names: manual lymphatic drainage; compression; exercise
  Groups: With lymphedema undergoing complete decongestive therapy (CDT)
Other: Standard imaging protocol — The standard imaging protocol entails noninvasive magnetic resonance imaging techniques including sodium and lymphatic angiography.

SUMMARY:
Recent evidence supports lymphatic regulation of tissue sodium handling, however fundamental gaps persist in knowledge regarding the role of lymphatics in human diseases of sodium dysregulation. The goal of this work is to apply novel, noninvasive imaging tools to measure relationships between lymphatic function and tissue sodium in patients with well-characterized lymphedema. Findings are intended to inform mechanisms of lymphatic clearance of tissue sodium, and provide novel imaging biomarkers of lymphedema progression and treatment response.

DETAILED DESCRIPTION:
The overall goal of this work is to apply and evaluate novel, noninvasive MRI technologies sensitive to sodium and lymphatic circulation in patients with well-characterized lymphatic disease. The results will clarify mechanisms of lymphatic clearance of tissue sodium, and evaluate novel biomarkers of lymphedema risk, progression, and treatment response. Recent evidence supports that lymphatics regulate interstitial sodium levels. When lymphatic clearance is impaired, hypertonic interstitial sodium results in tissue swelling, skin sodium storage, and poor blood pressure control. When lymphatic clearance is impaired in rodent models of lymphedema, lymph stasis and inflammation ensue, leading to tissue remodeling and fibrosis. These data suggest, but do not confirm, that impaired lymphatic clearance contributes to tissue sodium storage and fibrosis. However, this possibility has not been investigated rigorously owing to a lack of clinically-feasible measurement tools sensitive to sodium and lymphatics in humans. To address these gaps in knowledge, the investigators have developed a noninvasive MR lymphangiography (MRL) approach to quantify lymphatic vasculature in patients with unilateral lymphedema of the upper-extremities. They confirmed lateralized lymph stasis and enlarged lymphatic collector cross-sectional area that reduced following manual lymphatic drainage therapy. In parallel to these studies, the investigators optimized noninvasive sodium 23Na MRI for measurement of tissue sodium content (TSC) in the legs of patients with lymphatic insufficiency due to lipedema. In preliminary data, they demonstrate these methods together for the first time in patients with cancer-related lower-extremity lymphedema (LEL) who display significantly elevated skin TSC compared to controls (24.2±6.8 vs. 14.2±1.8 mmol/L, p<0.001, effect size Cohen's d=1.2). Evidence of lymphatic impairment on MRL and tissue sodium deposition are differential in patients with increasing disease severity, and modified by lymphatic complete decongestive therapy (CDT), motivating the following hypotheses:

Hypothesis (1): Skin TSC inversely correlates with lymphatic flow velocity; lymphatic flow velocity reduces and TSC increases following LN removal in patients at risk for lymphedema. Hypothesis (2): Skin TSC positively correlates with lymphedema stage; subcutaneous sodium co-localizes with fibrotic tissue in patients with lymphedema and fibrosis. Hypothesis (3): Skin TSC decreases and lymphatic flow velocity increases after CDT in affected limbs with LEL; imaging metrics are reproducible in healthy volunteers. Impact: Results will demonstrate relationships between tissue sodium and lymphatic dysfunction in human disease using noninvasive MRI technologies. This will outline clinically-feasible biomarkers of lymphedema risk, progression, and treatment response which could have significance for future clinical trials that seek to evaluate the impact of emerging lymphatic therapies on tissue sodium storage.

ELIGIBILITY:
Inclusion Criteria:

* Biologically Female
* Age range = 18-80 years
* BMI range = 18 to 40 kg/m2

Exclusion Criteria:

* Primary lymphedema
* Contraindication to 3T MRI
* Pregnant
* Severe claustrophobia
* Inability to provide written, informed consent
* Active infection anywhere in the body, or open wound on the lower-extremities or at locations for measurement
* Subjects who cannot adhere to the experimental protocols for any reason

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit adults who are at-risk for lower-extremity lymphedema (n=30) or who have lower-extremity secondary lymphedema (n=45).
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of tissue sodium content | Baseline to completion of routine course of physical therapy (approximately 6 weeks)
  Research participants will undergo periodic noninvasive sodium MRI after clinically-indicated complete decongestive therapy. The study team will measure change in tissue sodium content (mmol/L) in the treated extremities to study effects of lymphatic stimulation on sodium clearance.
Number of participants that changed lymphedema severity | Baseline to completion of routine course of physical therapy (approximately 6 weeks)
  Research participants will undergo periodic noninvasive magnetic resonance lymphangiography after clinically-indicated complete decongestive therapy. The study team will measure change in quantified lymphatic stasis in the treated extremities to study effects of lymphatic stimulation on lymphedema severity.
Concentration of tissue sodium content baseline | Baseline
  For participants at-risk or with lymphedema, noninvasive sodium MRI will measure tissue sodium content (mmol/L) in the extremities to study sodium in lymphedema.
Quantification of lymphatic states in extremities at baseline | Baseline
  For participants at-risk or with lymphedema, noninvasive MR lymphangiography will measure quantified lymphatic stasis in the extremities to study lymphatic physiology in lymphedema.

SECONDARY OUTCOMES:
Concentration in limb extracellular water | Baseline and after a routine course of physical therapy (approximately 6 weeks)
  Research participants will undergo periodic assessment by bioimpedance spectroscopy to estimate limb extracellular water (whole-limb resistance, Ohms) after clinically-indicated complete decongestive therapy. The study team will measure change in limb extracellular water (whole-limb resistance, Ohms) in the treated extremities to study effects of lymphatic stimulation on tissue composition.
Concentration in skin water | Baseline and after a routine course of physical therapy (approximately 6 weeks)
  Research participants will undergo periodic assessment by tissue dielectric probe to estimate skin water (% water) after clinically-indicated complete decongestive therapy. The study team will measure change in skin water (% water) in the treated extremities to study effects of lymphatic stimulation on tissue composition.
Change in skin elasticity | Baseline and after a routine course of physical therapy (approximately 6 weeks)
  Research participants will undergo periodic assessment by fibrometer probe to estimate skin elasticity (Newtons of induration) after clinically-indicated complete decongestive therapy. The study team will measure change in skin elasticity (Newtons of induration) in the treated extremities to study effects of lymphatic stimulation on tissue composition.
Concentration of limb extracellular water at baseline | Baseline
  For participants at-risk or with lymphedema, baseline limb extracellular water (whole-limb resistance, Ohms) will be estimated in the extremities to study tissue composition in lymphedema.
Baseline skin water | Baseline
  For participants at-risk or with lymphedema, baseline skin water (% water) will be estimated in the extremities to study tissue composition in lymphedema.
Baseline skin elasticity | Baseline
  For participants at-risk or with lymphedema, baseline skin elasticity (Newtons of induration) will be estimated in the extremities to study tissue composition in lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Rachelle Crescenzi, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided